CLINICAL TRIAL: NCT04992741
Title: The Effect of Health belıef Model Based educatıon and motıvatıonal intervıewıng on Mothers' Knowledge, belıef and attıtudes Towards Hpv vaccıne
Brief Title: Health Belief Model-based Education and Motivational Interview Regarding the HPV Vaccination Decision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin ATEŞEYAN (Other)
Responsible Party: Sponsor-Investigator, Yasemin ATEŞEYAN, lecturer, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YASEMIN-001
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: HPV VACCINATION
Keywords: HPV, Health Belief Model, Motivational Interview, Nursing
MeSH Terms: conditions — Papillomavirus Infections | interventions — Educational Status; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Masking Description: The two high schools included in the research will be determined as experimental and control groups by lottery method. By an independent researcher who was not involved in the study, 27 mothers from both schools who agreed to participate in the study will be selected by lottery method. Selected mothers will be called one by one by phone to be informed about the research, and the "Informed Consent Form" will be filled in via whatsapp and survey/scale forms will be applied. Participants will be blinded. The researcher (YA) cannot be blinded due to the nature of the research. When the research is completed, the data will be transferred to the computer environment by an independent researcher who does not know the A and B groups and the data will be analyzed by a statistician and the findings will be reported
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Health Belief Model Based Motivational Interview Group The application will be made by the researcher who has been trained in motivational interviewing techniques. Motivational interviews based on Health Belief Model will be made by telephone to mothers who have daughters studying in high school. There will be 3 interviews with mothers based on the benefits, barriers, sensitivity and severity perception structures of the Health Belief Model regarding HPV infection and vaccination, and each interview will last 15-20 minutes. One week after each interview, the questionnaire/scale forms will be sent via whatsapp and applied.
  Interventions: Other: education and motivational interview
- other (No Intervention): The control group will remain subject to the routine process without any intervention.

INTERVENTIONS:
Other: education and motivational interview — The control group will remain subject to the routine process without any intervention.
  Arms: Experimental

SUMMARY:
This research is a single-blind, randomized, parallel-controlled experimental study designed to determine the effect of Health Belief Model (SIM)-based motivational interviews given to mothers of high school students on mothers' knowledge, beliefs and attitudes towards HPV vaccine. . The hypotheses of the research; The experimental group that received training and motivational interviews within the framework of SIM had higher knowledge and perception of HPV infection and vaccination in the posttest than the control group that did not receive any application.

DETAILED DESCRIPTION:
Methods: In order to determine the sample size of the study, it was planned to work with a total of 54 patients, at least 27 patients in each group, in the power analysis performed by taking the reference information of the statistician and previous studies, and the study was completed with a total of 63 people (31 in the experimental group, 32 in the control group). The Health Belief Model-based motivational interview will be conducted over the phone and will last 15-20 minutes. One week after each motivational interview, a questionnaire and scale form will be applied to the mothers. After the third meeting, the study will be completed by applying the questionnaire and scale forms. Finally, the questionnaire for measurement will be filled and the research will be completed.

The control group will be subjected to routine processing without any intervention. Questionnaire forms were applied to the control group simultaneously with the experimental group. At the end of the study, a single-session motivational interview will be held by the researcher, since the patients in the control group have equal ethical rights. The primary result expected from the study is that mothers' perceptions of the benefit, sensitivity and severity of HPV vaccine increase, and their perception of barriers decreases. The secondary result expected from the study is the increase in mothers' knowledge about HPV infection and vaccination. The tertiary expected outcome of the study is that the mother sees her daughter at risk of HPV infection and decides to have her daughter vaccinated against HPV.

ELIGIBILITY:
Inclusion Criteria:

1. Those who live in Mersin and are female students in two high schools determined between 15.03.2020 and 15.06.2021.,
2. Daughter not vaccinated against HPV,
3. Undecided about getting her daughter vaccinated against HPV,
4. Who doesn't plan to have their daughter vaccinated against HPV,
5. who agreed to participate in the research,
6. Literate,
7. Can speak Turkish,,
8. Having no hearing or sight impairment that will prevent communication,,
9. Able to talk on the phone and use whatsapp,,
10. Participants without a diagnosed psychiatric problem were included in the study..

Exclusion Criteria:

1. Having her daughter vaccinated against HPV,
2. Thinking of getting her daughter vaccinated against HPV,
3. Who refused to participate in the research,
4. Illiterate,
5. Don't speak Turkish,
6. People with hearing or sight impairments that may interfere with communication,
7. Can't talk on the phone and can't use whatsapp,
8. Participants with diagnosed psychiatric problems were excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures: Health Belief was assessed with the Health Belief Model Scale for Human Papilloma Virus Infection and Vaccination | Change from before implementation, 1th week, 2th week and 3th week of practice
  It was developed by Kim (2012) to measure health beliefs towards the HPV vaccine. The scale consists of 4 subscales: benefits (1-3 items), perceived disability (10-14 items), sensitivity (4-5 items), severity (6-9 items) and a total of 14 items. The scale items are interpreted as four-point likert type, with 1 as "not at all", 2 as "a little", 3 as "quite a lot", and 4 as "a lot". The total score range of the scale is 14-56. As the scale score increases, the perception also increases.
HPV information assessed with HPV information scale | Change from before implementation, Change from before implementation, 1th week, 2th week and 3th week of practice
  The HPV knowledge scale was developed by Waller et al (2013) to measure the knowledge levels of individuals about HPV, HPV vaccine and screening tests. In the scale with a total of 33 items; It consists of four sub-dimensions: general HPV information (1-16 items), HPV screening test information (17-22 items), general HPV vaccine information (23-27 items) and information about the current HPV vaccination program (28-33 items). Participants are expected to mark each item of the scale as "Yes", "No" and "I don't know". In the evaluation phase, each correct answer is scored with=1, while incorrect answers and I don't know are scored with=0. In order to avoid bias in the answers, the correct and incorrect answers were mixed as in the original scale. The total score to be obtained from the scale is between 0-33, and a high score indicates a high level of knowledge about HPV, HPV screening tests and HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Ateşeyan, Study Chair — Turkey, Mersin University, Mersin, Yenişehir, Turkey, 33343
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Derived] Ateseyan Y, Gungormus Z. Web and theory-based motivational interviews in encouraging mothers for HPV vaccination of their daughters: A randomized controlled study. J Pediatr Nurs. 2024 Sep-Oct;78:e279-e288. doi: 10.1016/j.pedn.2024.07.016. Epub 2024 Jul 26. PMID 39060172